CLINICAL TRIAL: NCT06866522
Title: Light Reflection on Human Skin in Whole-Body Photobiomodulation Therapy: Clinical Trial
Brief Title: Light Reflection on Human Skin in Whole-Body Photobiomodulation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Lara Maria Bataglia Espósito, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 70368823.8.0000.5504; 2023/07857-6 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2025-02-28; First posted 2025-03-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Photobiomodulation Therapy; Phototype
Keywords: photobiomodulation; low-level laser therapy; skin optics; melanin; light reflection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photobiomodulation Reflection Group (Experimental): This group received measures of the light reflection using a whole-body photobiomodulation therapy with a Joovv device. In this group, participants were subclassified with the Fitzpatrick scale for their phototypes.
  Interventions: Device: Whole-body Photobiomodulation Therapy

INTERVENTIONS:
Device: Whole-body Photobiomodulation Therapy — Whole-body Photobiomodulation Therapy applied for approximately 10 minutes, being 5 minutes with the red wavelength and 5 minutes with the infrared wavelength.

SUMMARY:
Photobiomodulation therapy (PBMT) is based on exposing biological tissues to low-intensity light, with effects depending on the light-tissue interaction. When irradiated without skin contact, part of the incident light is reflected and lost. In this context, the amount of reflected light in PBMT applied without skin contact, as well as the influence of skin phototype, has not yet been established. Objective: To quantify the reflection of light from PBMT on the skin of men and women aged 18 to 30 years, considering skin phototypes. Methodology: Participants will be divided into three groups based on skin phototype (Group 1: phototypes I and II; Group 2: phototypes III and IV; Group 3: phototypes V and VI) and sex. They will be subjected to whole-body PBMT with red light (660 nm; 31.85±3.85 mW; 45.50±5.07 mW/cm²) and infrared light (850 nm; 25.29±2.99 mW; 36.13±4.27 mW/cm²) at 20 cm from the light-emitting source, with measurement of light reflection in the regions of the brachial biceps, abdomen, lumbar, anterior and posterior thigh, and calf using a power and energy analyzer (powermeter PM100D and sensor S130C, 0.7 cm²). Data will be analyzed for normality and groups were compared with a significance level of 5%

ELIGIBILITY:
Inclusion Criteria:

* male and female
* age between 18 and 30 years
* body mass index (BMI) between 18.5 and 29.9 kg/m2.

Exclusion Criteria:

* tattoo in the light reflection assessment areas
* history of skin cancer
* skin lesions such as open wounds in the mid-thigh, abdomen, biceps brachii, back and calf
* patients with cognitive difficulty reporting thermal sensation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Light Reflection | Acute measurement. The measurement will be performed just during the light therapy irradiation, on the day of the procedure.
  Light reflection will be measured in mW with a PowerMeter Device in the angles of 30º, 60º and 90º considering the participant in front of the whole-body photobiomodulation therapy device.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Carlos (UFSCar), São Carlos, São Paulo, Brazil